CLINICAL TRIAL: NCT04132336
Title: A Randomized, Double-Blind, Single-Dose, Parallel, Placebo-Controlled Trial to Determine the Dose of Caffeine in a Fixed Dose Combination Tablet of Naproxen Sodium and Caffeine to Effectively Alleviate Postsurgical Dental Pain
Brief Title: Study to Find Out the Optimal Dose of Caffeine in the Combination Tablet of Naproxen Sodium and Caffeine in Patients Experiencing Moderate to Severe Pain After Having Wisdom Teeth Removed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21069; 2019-003513-33 (EudraCT Number)
Record Dates: First submitted 2019-10-08; First posted 2019-10-18 (Actual); Results first posted 2021-06-16 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Pain, Postoperative
Keywords: Dental pain
MeSH Terms: conditions — Pain, Postoperative; Toothache | interventions — Naproxen; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Naproxen sodium/caffeine - Dose 1 (Experimental): Participants received a single dose of two tablets of naproxen sodium/caffeine (low dose/medium low dose) after extraction of third molars
  Interventions: Drug: Naproxen sodium/Caffeine (BAY2880376)
- Naproxen sodium/caffeine - Dose 2 (Experimental): Participants received a single dose of two tablets of naproxen sodium/caffeine (low dose/low dose) after extraction of third molars
  Interventions: Drug: Naproxen sodium/Caffeine (BAY2880376)
- Naproxen sodium/caffeine - Dose 3 (Experimental): Participants received a single dose of one tablet of naproxen sodium/caffeine (low dose/ medium low dose) plus one tablet of placebo after extraction of third molars
  Interventions: Drug: Naproxen sodium/Caffeine (BAY2880376)
- Naproxen sodium/caffeine - Dose 4 (Experimental): Participants received a single dose of one tablet of naproxen sodium/caffeine (low dose/ low dose) plus one tablet of placebo after extraction of third molars
  Interventions: Drug: Naproxen sodium/Caffeine (BAY2880376)
- Naproxen sodium (Active Comparator): Participants received a single dose of one tablet of naproxen sodium (low dose) plus one tablet of placebo after extraction of third molars
  Interventions: Drug: Naproxen sodium (Aleve)
- Caffeine (Active Comparator): Participants received a single dose of two tablets of caffeine (medium low dose) after extraction of third molars
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator): Participants received a single dose of two tablets of matching placebo after extraction of third molars
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen sodium/Caffeine (BAY2880376) — Tablet, oral, single dose
  Arms: Naproxen sodium/caffeine - Dose 1; Naproxen sodium/caffeine - Dose 2; Naproxen sodium/caffeine - Dose 3; Naproxen sodium/caffeine - Dose 4
Drug: Naproxen sodium (Aleve) — Tablet, oral, single dose
  Arms: Naproxen sodium
Drug: Caffeine — Tablet, oral, single dose
  Arms: Caffeine
Drug: Placebo — Tablet, oral, single dose
  Arms: Placebo

SUMMARY:
The researchers in this study wanted to find out the optimal dose of Caffeine in the combination tablet of Naproxen Sodium and Caffeine that works in patients experiencing moderate to severe pain after having wisdom teeth removed. In the US, Naproxen has been marketed since 1976, and Naproxen Sodium has been approved for over-the-counter (OTC) use since 1994 for the temporary relief of minor aches and pains. Caffeine, which is generally consumed as coffee, tea or cocoa, has been shown to enhance the effectiveness of various pain relievers, and therefore is accepted as an additive to painkillers like aspirin and acetaminophen. Patients participating in this study underwent a surgery to remove 3 or 4 wisdom teeth. If the pain severity after the surgery met the study requirement, patients would receive oral tablet(s) of Naproxen Sodium and Caffeine, or Naproxen Sodium, or Caffeine, or placebo (drug with no active ingredient). Patients could also receive additional pain medication when needed. Researchers would also learn if the patients have any medical problems during the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male or female volunteers 16 years of age or older;
* Body mass index (BMI) 18.5 to 35.0 kg/m^2 inclusive as measured by the National Institutes of Health (NIH) BMI Calculator;
* Participants will undergo surgical extraction of three or four third molars, two of which must be mandibular molars. Maxillary third molars may be removed regardless of impaction level. The mandibular extractions must have a trauma rating of mild or moderate and meet one of the following scenarios: two full bony impactions; two partial bony impactions; one full bony impaction in combination with one partial bony impaction. supernumerary teeth present may also be removed at the discretion of the oral surgeon;
* Have not taken any form of medication, nutritional supplements with analgesic properties (e.g. gamma-Aminobutyric acid [GABA], turmeric) or herbal supplements (i.e., St. John's Wort) within 5 days of admission (except for oral contraceptives, prophylactic antibiotics, multivitamin supplements, or other routine medications to treat benign conditions (such as antibiotics to treat acne), and agree not to take any medication (other than that provided to them) throughout the study;
* Use of only short-acting local anesthetic (e.g., mepivacaine or lidocaine) preoperatively, with or without a vasoconstrictor and nitrous oxide at the discretion of the Investigator;
* Have moderate to severe postoperative pain on the Categorical Pain Intensity Scale (a score of at least 2 on a 4 point scale) and a score of ≥ 5 on the 0-10 pain intensity Numerical Rating Scale (NRS) within 4.5 hours post-surgery.

Exclusion Criteria:

* History of hypersensitivity to naproxen sodium, caffeine, ibuprofen, nonsteroidal anti-inflammatory drug (NSAIDS), aspirin, similar pharmacological agents, local anesthetics, rescue medication or components of the investigational products;
* Evidence or history of clinically significant (in the judgment of the investigator) hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including hypertension and cardiac arrhythmia), hepatic, psychiatric, neurologic diseases, or malignancies within the last 5 years;
* Participants with the following medical conditions may be eligible at the discretion of the investigator: attention deficit hyperactivity disorder (ADHD) on a stable dose regimen of methylphenidate/(dextro) amphetamine for at least 6 months; participants with hypothyroidism on a stable dose of synthetic thyroid hormone for at least 6 months;
* Have received any form of treatment in the form of medication for depression in the past 6 months or any form of psychotropic agent (including selective serotonin uptake inhibitors [SSRI] but excluding ADHD medications described above) within the last 6 months;
* Relevant concomitant disease such as asthma (exercise induced asthma is permitted);
* Current or past history of gastrointestinal ulceration, gastrointestinal bleeding or other bleeding disorder(s);
* Acute illness or active local infection prior to surgery that can interfere with the conduct of the study in the judgment of the investigator;
* Use of any over-the-counter (OTC) or prescription medications with which the administration of naproxen, acetaminophen, ibuprofen, any other NSAID, (e.g., tramadol) or if a medication is contraindicated;
* Use of any medications within 5 days of surgery until discharge from the study site (except oral contraceptives, prophylactic antibiotics, synthetic thyroid hormones, methylphenidate or medications to treat benign conditions such as antibiotics to treat acne);
* Use of caffeine within 2 days prior to the study;
* Habits of high consumption of caffeine (>400 mg/day equivalent to about 3-4 cups of coffee per day);
* Habituation to analgesic drugs including opioids (i.e., routine use of oral analgesics 5 or more times per week for greater than 3 weeks within the past 2 years);
* Surgeon's trauma rating of severe following surgery.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- JBR Clinical Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at a single center in United States with first participant first visit on 12-Nov-2019 and last participant last visit on 02-Mar-2020. Study was completed on 03-Mar-2020 (End of follow up, phone call).
Pre-assignment Details: A total of 193 participants, including 32 in each of the naproxen sodium containing groups, 16 in the caffeine group, and 17 in the placebo group, underwent dental surgery and were randomized to study drug
Groups:
- Naproxen Sodium/Caffeine-Dose 1: Participants received a single dose of two tablets of naproxen sodium/caffeine (low dose/medium low dose) after extraction of third molars
- Naproxen Sodium/Caffeine-Dose 2: Participants received a single dose of two tablets of naproxen sodium/caffeine (low dose/low dose) after extraction of third molars
- Naproxen Sodium/Caffeine-Dose 3: Participants received a single dose of one tablet of naproxen sodium/caffeine (low dose/ medium low dose) plus one tablet of placebo after extraction of third molars
- Naproxen Sodium/Caffeine-Dose 4: Participants received a single dose of one tablet of naproxen sodium/caffeine (low dose/ low dose) plus one tablet of placebo after extraction of third molars
Period: Overall Study
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Started | 32 | 32 | 32 | 32 | 32 | 16 | 17
Completed | 32 | 31 | 32 | 32 | 32 | 16 | 17
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo | Total
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 16 | 17 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.0 (1.03) | 17.4 (2.42) | 17.1 (1.34) | 17.3 (1.49) | 17.9 (2.74) | 17.3 (1.70) | 17.7 (1.40) | 17.4 (1.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 16 | 10 | 14 | 5 | 5 | 77
  Male | 19 | 18 | 16 | 22 | 18 | 11 | 12 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 3 | 2 | 3 | 0 | 10
  Not Hispanic or Latino | 30 | 32 | 32 | 29 | 30 | 13 | 17 | 183
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Baseline Pain Intensity Score [Count of Participants; unit: Participants]
  No Pain (0) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mild Pain (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Moderate Pain (2) | 15 | 13 | 12 | 11 | 11 | 3 | 5 | 70
  Severe Pain (3) | 17 | 19 | 20 | 21 | 21 | 13 | 12 | 123

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPID) Over 8 Hours
Description: Pain intensity is measured using Numerical Rating Scale (from 0 to 10: 0 = no pain, 10 = worst possible pain). For each post dose time point, pain intensity difference (PID) is derived by subtracting the pain intensity at the post dose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference is indicative of improvement. Sum of Pain Intensity Differences (SPIDs) was calculated by multiplying the PID score at each post-dose time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. SPID over 8 hours ranges from -80 to 80. A higher value indicates a better pain reduction.
Time Frame: Up to 8 hours post dose
Measure: Mean (Standard Deviation); unit: Scores on a scale*hours
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 32 | 16 | 16
Scores on a scale*hours | 35.45 (14.517) [lower limit 14.517] | 37.87 (16.876) [lower limit 16.876] | 30.70 (17.679) [lower limit 17.679] | 36.02 (14.825) [lower limit 14.825] | 29.95 (19.067) [lower limit 19.067] | 8.75 (21.465) [lower limit 21.465] | 6.03 (17.810) [lower limit 17.810]

2. Secondary Outcome: Sum of Pain Intensity Differences (SPIDs) From 0 to 2, 4 and 12 Hours Post-dose
Description: Pain intensity is measured using Numerical Rating Scale (from 0 to 10: 0 = no pain, 10 = worst possible pain). For each post dose time point, pain intensity difference (PID) is derived by subtracting the pain intensity at the post dose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference is indicative of improvement. Sum of Pain Intensity Differences (SPIDs) was calculated by multiplying the PID score at each post-dose time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. SPID 0-2 ranges from -20 to 20, SPID 0-4 ranges from -40 to 40 and SPID 0-12 ranges from -120 to 120. A higher value indicates a better pain reduction.
Time Frame: Up to 2 hours, 4 hours and 12 hours post dose
Measure: Mean (Standard Deviation); unit: Scores on a scale*hours
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 32 | 16 | 16
Scores on a scale*hours
  SPID 0-2 | 8.30 (3.141) [lower limit 3.141] | 8.68 (3.789) [lower limit 3.789] | 7.17 (3.721) [lower limit 3.721] | 6.92 (3.501) [lower limit 3.501] | 6.05 (3.511) [lower limit 3.511] | 2.13 (4.060) [lower limit 4.060] | 1.16 (2.925) [lower limit 2.925]
  SPID 0-4 | 18.02 (6.387) [lower limit 6.387] | 19.26 (8.019) [lower limit 8.019] | 15.58 (7.697) [lower limit 7.697] | 17.05 (7.232) [lower limit 7.232] | 14.33 (8.391) [lower limit 8.391] | 4.50 (9.604) [lower limit 9.604] | 2.59 (7.625) [lower limit 7.625]
  SPID 0-12 | 50.58 (24.237) [lower limit 24.237] | 52.45 (27.305) [lower limit 27.305] | 44.80 (28.929) [lower limit 28.929] | 52.45 (23.022) [lower limit 23.022] | 43.08 (30.034) [lower limit 30.034] | 12.44 (32.059) [lower limit 32.059] | 1.15 (2.833) [lower limit 2.833]

3. Secondary Outcome: Total Pain Relief (TOTPAR) Over 8 Hours
Description: Pain relief is measured using Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief). Total Pain Relief is calculated as the area under the curve of pain relief score over time for the given time period by multiplying the pain relief score at each time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. TOTPAR over 8 hours ranges from 0 to 32, a higher value indicates more pain relief.
Time Frame: Up to 8 hours post dose
Measure: Mean (Standard Deviation); unit: Scores on a scale*hours
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 32 | 16 | 16
Scores on a scale*hours | 19.58 (7.007) [lower limit 7.007] | 20.26 (7.673) [lower limit 7.673] | 17.41 (8.063) [lower limit 8.063] | 19.53 (6.448) [lower limit 6.448] | 16.27 (8.514) [lower limit 8.514] | 7.03 (9.283) [lower limit 9.283] | 5.44 (7.709) [lower limit 7.709]

4. Secondary Outcome: Total Pain Relief (TOTPAR) From 0 to 2, 4 and 12 Hours Post-dose
Description: Pain relief is measured using Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief). Total Pain Relief is calculated as the area under the curve of pain relief score over time for the given time period by multiplying the pain relief score at each time point by the duration (in hours) since the preceding time point and then summing these values over the specific time period. TOTPAR 0-2 ranges from 0 to 8, TOTPAR 0-4 ranges from 0 to 16, and TOTPAR 0-12 ranges from 0 to 48. A higher value indicates more pain relief
Time Frame: Up to 2 hours, 4 hours and 12 hours post dose
Measure: Mean (Standard Deviation); unit: Scores on a scale*hours
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 32 | 16 | 16
Scores on a scale*hours
  TOTPAR 0-2 | 4.83 (1.401) [lower limit 1.401] | 4.77 (1.731) [lower limit 1.731] | 4.22 (1.596) [lower limit 1.596] | 3.97 (1.436) [lower limit 1.436] | 3.52 (1.644) [lower limit 1.644] | 1.66 (1.767) [lower limit 1.767] | 1.06 (1.328) [lower limit 1.328]
  TOTPAR 0-4 | 10.27 (2.750) [lower limit 2.750] | 10.29 (3.449) [lower limit 3.449] | 8.84 (3.286) [lower limit 3.286] | 9.28 (2.842) [lower limit 2.842] | 7.86 (3.813) [lower limit 3.813] | 3.59 (4.148) [lower limit 4.148] | 2.44 (3.281) [lower limit 3.281]
  TOTPAR 0-12 | 28.20 (12.262) [lower limit 12.262] | 28.26 (12.690) [lower limit 12.690] | 25.13 (13.291) [lower limit 13.291] | 28.72 (10.678) [lower limit 10.678] | 22.95 (13.206) [lower limit 13.206] | 10.28 (13.882) [lower limit 13.882] | 8.44 (12.419) [lower limit 12.419]

5. Secondary Outcome: Time to First Use of Rescue Medication
Time Frame: Up to 12 hours post dose
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 32 | 16 | 16
hours | NA [NA to NA] — NA= insufficient number of participants with events | NA [8.967 to NA] — NA= insufficient number of participants with events | NA [8.817 to NA] — NA= insufficient number of participants with events | NA [NA to NA] — NA= insufficient number of participants with events | NA [8.125 to NA] — NA= insufficient number of participants with events | 2.083 [1.275 to NA] — NA= insufficient number of participants with events | 2.125 [1.408 to NA] — NA= insufficient number of participants with events

6. Secondary Outcome: The Cumulative Percentage of Participants Taking Rescue Medication
Time Frame: Up to 12 hours post dose
Measure: Number; unit: Percentage of participants
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 32 | 16 | 16
Percentage of participants
  0.5 Hours Post-Dose | 0 | 0 | 0 | 0 | 0 | 0 | 0
  1 Hour Post-Dose | 0 | 0 | 0 | 0 | 0 | 0 | 0
  1.5 Hours Post-Dose | 0 | 3.2 | 3.1 | 0 | 0 | 37.5 | 25.0
  2 Hours Post-Dose | 0 | 3.2 | 3.1 | 0 | 0 | 50 | 37.5
  3 Hours Post-Dose | 0 | 6.5 | 6.3 | 3.1 | 15.6 | 56.3 | 56.3
  4 Hours Post-Dose | 3.1 | 6.5 | 9.4 | 3.1 | 18.8 | 56.3 | 68.8
  5 Hours Post-Dose | 9.4 | 6.5 | 15.6 | 3.1 | 18.8 | 62.5 | 68.8
  6 Hours Post-Dose | 9.4 | 9.7 | 18.8 | 6.3 | 21.9 | 68.8 | 68.8
  7 Hours Post-Dose | 12.5 | 9.7 | 21.9 | 6.3 | 21.9 | 68.8 | 68.8
  8 Hours Post-Dose | 15.6 | 9.7 | 21.9 | 9.4 | 21.9 | 68.8 | 75.0
  9 Hours Post-Dose | 21.9 | 25.8 | 25.0 | 9.4 | 28.1 | 68.8 | 75.0
  10 Hours Post-Dose | 25.0 | 25.8 | 28.1 | 15.6 | 31.3 | 68.8 | 75.0
  11 Hours Post-Dose | 25.0 | 25.8 | 28.1 | 15.6 | 34.4 | 68.8 | 75.0
  12 Hours Post-Dose | 25.0 | 29.0 | 28.1 | 18.8 | 34.4 | 75.0 | 75.0

7. Secondary Outcome: Pain Intensity Difference (PID) at Each Evaluation
Description: Pain intensity is measured using Numerical Rating Scale (from 0 to 10: 0 = no pain, 10 = worst possible pain). For each post dose time point, pain intensity difference (PID) is derived by subtracting the pain intensity at the post dose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference is indicative of improvement
Time Frame: Up to 12 hours post dose
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 31 | 32 | 31 | 32 | 16 | 16
Scores on a scale
  0.5 Hours Post-Dose | 2.3 (2.07) | 2.6 (1.82) | 2.1 (2.23) | 1.4 (1.56) | 1.5 (1.34) | 0.8 (0.98) | 0.5 (0.89)
  1 Hour Post-Dose | 4.2 (1.88) | 4.2 (2.44) | 3.7 (1.95) | 3.4 (2.39) | 2.9 (1.88) | 1.2 (2.26) | 0.6 (1.71)
  1.5 Hours Post-Dose | 4.9 (1.67) | 5.1 (2.26) | 4.3 (1.98) | 4.2 (2.32) | 3.7 (2.16) | 1.2 (2.79) | 0.7 (1.74)
  2 Hours Post-Dose | 5.1 (1.76) | 5.5 (2.20) | 4.3 (2.23) | 4.8 (2.23) | 4.1 (2.22) | 1.1 (2.67) | 0.5 (1)
  3 Hours Post-Dose | 5.0 (1.82) | 5.4 (2.27) | 4.3 (2.33) | 5.0 (2.29) | 4.0 (2.83) | 1.1 (2.85) | 0.6 (2.42)
  4 Hours Post-Dose | 4.8 (2.17) | 5.2 (2.59) | 4.1 (2.62) | 5.1 (2.27) | 4.3 (2.82) | 1.3 (3.11) | 0.9 (2.78)
  5 Hours Post-Dose | 4.7 (2.28) | 5.0 (2.42) | 4.0 (2.72) | 5.0 (2.25) | 4.1 (2.83) | 1.1 (3.14) | 1.0 (2.92)
  6 Hours Post-Dose | 4.6 (2.24) | 4.8 (2.42) | 3.8 (2.87) | 4.9 (2.40) | 3.9 (2.88) | 1.1 (3.19) | 1.0 (3.06)
  7 Hours Post-Dose | 4.3 (2.55) | 4.5 (2.45) | 3.8 (3.07) | 4.7 (2.31) | 3.9 (3.08) | 1.1 (3.36) | 0.8 (2.49)
  8 Hours Post-Dose | 4.0 (2.53) | 4.2 (2.65) | 3.7 (3.12) | 4.3 (2.29) | 3.7 (2.96) | 0.9 (2.95) | 0.7 (2.65)
  9 Hours Post-Dose | 3.8 (2.71) | 3.8 (3.12) | 3.6 (3.00) | 4.2 (2.45) | 3.6 (3.14) | 1.1 (3.09) | 0.8 (2.74)
  10 Hours Post-Dose | 3.8 (2.88) | 3.7 (3.04) | 3.4 (3.15) | 4.1 (2.60) | 3.3 (3.07) | 1.1 (3.07) | 0.9 (2.99)
  11 Hours Post-Dose | 3.8 (2.92) | 3.5 (3.02) | 3.6 (3.17) | 4.2 (2.79) | 3.1 (3.02) | 0.8 (2.99) | 0.9 (2.96)
  12 Hours Post-Dose | 3.8 (2.97) | 3.6 (3.06) | 3.5 (3.38) | 4.0 (2.92) | 3.1 (2.97) | 0.8 (3.00) | 0.9 (2.96)

8. Secondary Outcome: Peak Pain Intensity Difference (PID)
Description: Pain intensity is measured using Numerical Rating Scale (from 0 to 10: 0 = no pain, 10 = worst possible pain). Participants circle a number (from 0 to 10) on the Numerical Rating Scale to indicate the severity the pain they are experiencing at baseline and at each post dose time point. For each post dose time point, pain intensity difference (PID) is derived by subtracting the pain intensity at the post dose time point from the baseline intensity score (baseline score - post-baseline score).
Time Frame: Up to 12 hours post dose
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 32 | 16 | 16
Scores on a scale | 6.0 (1.53) [lower limit 1.53] | 6.2 (1.97) [lower limit 1.97] | 5.9 (2.01) [lower limit 2.01] | 6.3 (1.72) [lower limit 1.72] | 5.3 (2.57) [lower limit 2.57] | 2.7 (2.94) [lower limit 2.94] | 2.3 (2.98) [lower limit 2.98]

9. Secondary Outcome: Pain Relief Score at Each Evaluation
Description: Pain relief is measured using Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief)
Time Frame: Up to 12 hours post dose
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 32 | 16 | 16
Scores on a scale
  0.5 Hours Post-Dose | 1.6 (1.08) [lower limit 1.08] | 1.5 (0.89) [lower limit 0.89] | 1.5 (1.02) [lower limit 1.02] | 0.9 (0.80) [lower limit 0.80] | 1.0 (0.74) [lower limit 0.74] | 0.6 (0.62) [lower limit 0.62] | 0.4 (0.63) [lower limit 0.63]
  1 Hours Post-Dose | 2.4 (0.84) [lower limit 0.84] | 2.3 (1.22) [lower limit 1.22] | 2.2 (0.91) [lower limit 0.91] | 2.0 (1.14) [lower limit 1.14] | 1.8 (0.91) [lower limit 0.91] | 0.9 (1.00) [lower limit 1.00] | 0.6 (0.81) [lower limit 0.81]
  1.5 Hours Post-Dose | 2.8 (0.64) [lower limit 0.64] | 2.8 (0.99) [lower limit 0.99] | 2.3 (0.87) [lower limit 0.87] | 2.4 (0.91) [lower limit 0.91] | 2.0 (1.05) [lower limit 1.05] | 0.9 (1.24) [lower limit 1.24] | 0.6 (0.73) [lower limit 0.73]
  2 Hours Post-Dose | 2.8 (0.85) [lower limit 0.85] | 2.9 (1.01) [lower limit 1.01] | 2.4 (1.01) [lower limit 1.01] | 2.6 (0.79) [lower limit 0.79] | 2.2 (1.01) [lower limit 1.01] | 0.8 (1.05) [lower limit 1.05] | 0.5 (0.82) [lower limit 0.82]
  3 Hours Post-Dose | 2.8 (0.79) [lower limit 0.79] | 2.8 (0.97) [lower limit 0.97] | 2.4 (1.04) [lower limit 1.04] | 2.6 (0.91) [lower limit 0.91] | 2.1 (1.21) [lower limit 1.21] | 0.9 (1.24) [lower limit 1.24] | 0.6 (1.09) [lower limit 1.09]
  4 Hours Post-Dose | 2.7 (1.07) [lower limit 1.07] | 2.7 (1.19) [lower limit 1.19] | 2.3 (1.16) [lower limit 1.16] | 2.7 (0.96) [lower limit 0.96] | 2.2 (1.26) [lower limit 1.26] | 1.0 (1.37) [lower limit 1.37] | 0.8 (1.18) [lower limit 1.18]
  5 Hours Post-Dose | 2.6 (1.16) [lower limit 1.16] | 2.6 (1.15) [lower limit 1.15] | 2.3 (1.27) [lower limit 1.27] | 2.7 (1.00) [lower limit 1.00] | 2.2 (1.24) [lower limit 1.24] | 0.9 (1.36) [lower limit 1.36] | 0.8 (1.18) [lower limit 1.18]
  6 Hours Post-Dose | 2.4 (1.16) [lower limit 1.16] | 2.6 (1.18) [lower limit 1.18] | 2.2 (1.35) [lower limit 1.35] | 2.7 (1.10) [lower limit 1.10] | 2.1 (1.30) [lower limit 1.30] | 0.9 (1.45) [lower limit 1.45] | 0.8 (1.24) [lower limit 1.24]
  7 Hours Post-Dose | 2.3 (1.34) [lower limit 1.34] | 2.5 (1.15) [lower limit 1.15] | 2.1 (1.38) [lower limit 1.38] | 2.5 (1.08) [lower limit 1.08] | 2.1 (1.29) [lower limit 1.29] | 0.9 (1.50) [lower limit 1.50] | 0.8 (1.28) [lower limit 1.28]
  8 Hours Post-Dose | 2.1 (1.33) [lower limit 1.33] | 2.3 (1.28) [lower limit 1.28] | 2.1 (1.46) [lower limit 1.46] | 2.4 (1.19) [lower limit 1.19] | 2.0 (1.28) [lower limit 1.28] | 0.8 (1.33) [lower limit 1.33] | 0.7 (1.25) [lower limit 1.25]
  9 Hours Post-Dose | 2.2 (1.40) [lower limit 1.40] | 2.1 (1.48) [lower limit 1.48] | 2.0 (1.45) [lower limit 1.45] | 2.3 (1.12) [lower limit 1.12] | 1.9 (1.41) [lower limit 1.41] | 0.9 (1.36) [lower limit 1.36] | 0.8 (1.34) [lower limit 1.34]
  10 Hours Post-Dose | 2.2 (1.51) [lower limit 1.51] | 2.0 (1.43) [lower limit 1.43] | 1.8 (1.42) [lower limit 1.42] | 2.3 (1.28) [lower limit 1.28] | 1.8 (1.41) [lower limit 1.41] | 0.9 (1.36) [lower limit 1.36] | 0.8 (1.34) [lower limit 1.34]
  11 Hours Post-Dose | 2.1 (1.52) [lower limit 1.52] | 1.9 (1.40) [lower limit 1.40] | 1.9 (1.48) [lower limit 1.48] | 2.4 (1.34) [lower limit 1.34] | 1.4 (1.32) [lower limit 1.32] | 0.8 (1.34) [lower limit 1.34] | 0.8 (1.34) [lower limit 1.34]
  12 Hours Post-Dose | 2.2 (1.55) [lower limit 1.55] | 1.9 (1.46) [lower limit 1.46] | 2.0 (1.51) [lower limit 1.51] | 2.2 (1.45) [lower limit 1.45] | 1.6 (1.39) [lower limit 1.39] | 0.8 (1.34) [lower limit 1.34] | 0.8 (1.34) [lower limit 1.34]

10. Secondary Outcome: Peak Pain Relief Score
Description: Pain relief is measured using Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief). At each post-dose time point, participants check the appropriate box (from 0 to 4) on the Categorical Pain Relief Rating Scale to indicate the relief from starting pain at the post dose time points.
Time Frame: Up to 12 hours post dose
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 32 | 16 | 16
Scores on a scale | 3.3 (0.62) [lower limit 0.62] | 3.2 (0.78) [lower limit 0.78] | 3.0 (0.82) [lower limit 0.82] | 3.1 (0.66) [lower limit 0.66] | 2.6 (1.01) [lower limit 1.01] | 1.6 (1.55) [lower limit 1.55] | 1.3 (1.39) [lower limit 1.39]

11. Secondary Outcome: Global Assessment of the Investigational Product
Description: Global assessment is performed either at 12 hours post-dose or immediately prior to the first intake of rescue medication. Global assessment is based on the question 'Overall, I would rate the study medication I received: 0=Poor, 1=Fair, 2=Good, 3=Very Good, 4=Excellent.'
Time Frame: Up to 12 hours post dose
Measure: Count of Participants; unit: Participants
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 31 | 32 | 32 | 32 | 16 | 16
Participants
  Poor (0) | 1 | 1 | 1 | 1 | 4 | 8 | 10
  Fair (1) | 2 | 1 | 4 | 2 | 5 | 1 | 2
  Good (2) | 5 | 6 | 9 | 7 | 6 | 4 | 1
  Very Good (3) | 18 | 14 | 13 | 17 | 14 | 2 | 3
  Excellent (4) | 6 | 9 | 5 | 5 | 3 | 1 | 0

12. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Up to 5 days post dose
Measure: Count of Participants; unit: Participants
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 16 | 17
Participants | 6 | 3 | 1 | 2 | 3 | 5 | 4

13. Secondary Outcome: The Number of Participants With Clinically Significant Changes in Physical Examinations and Vital Signs
Time Frame: Up to 5 days post dose
Measure: Count of Participants; unit: Participants
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 16 | 17
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 days post-dose
Arm/Group | Naproxen Sodium/Caffeine-Dose 1 | Naproxen Sodium/Caffeine-Dose 2 | Naproxen Sodium/Caffeine-Dose 3 | Naproxen Sodium/Caffeine-Dose 4 | Naproxen Sodium | Caffeine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32 | 0/32 | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32 | 0/32 | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 6/32 | 3/32 | 1/32 | 2/32 | 3/32 | 5/16 | 4/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium/Caffeine-Dose 1 (N=32) | Naproxen Sodium/Caffeine-Dose 2 (N=32) | Naproxen Sodium/Caffeine-Dose 3 (N=32) | Naproxen Sodium/Caffeine-Dose 4 (N=32) | Naproxen Sodium (N=32) | Caffeine (N=16) | Placebo (N=17)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 4 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alveolar osteitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Other pre-specified outcomes (non-key secondary) "Time to first perceptible relief/meaningful relief/perceptible relief confirmed by meaningful relief" and "Cumulative percentage of subjects with at least '2-point PID' over time" were also analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT04132336/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT04132336/SAP_001.pdf